CLINICAL TRIAL: NCT04480931
Title: Pilot Testing of a Mobile Health Intervention Designed to Increase Physical Activity and Improve Morbidity and Mortality-related Outcomes Among Pregnant and Postpartum Women in a Rural Setting
Brief Title: Pilot Testing a Mobile App to Designed to Increase Physical Activity Among Pregnant and Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Collaborators: University of Kentucky (Other)
Responsible Party: Principal Investigator, Rachel Tinius, Assistant Professor, Western Kentucky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-257
Record Dates: First submitted 2020-07-08; First posted 2020-07-22 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Pregnancy; Postpartum
Keywords: exercise; physical activity; mobile health; intervention
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Pregnant women will be recruited ~20 weeks pregnant and after baseline assessments, randomized into the control or intervention group. The intervention group will utilize the mhealth intervention, while the control group will receive basic educational materials only.
Masking Description: The participant (as well as the study team and the health care provider) will know after randomization whether or not they are being provided access to the mobile app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Intervention Group (Experimental): This group will be provided with the mobile health app (including introductory videos on how to use its features).
  Interventions: Behavioral: mHealth Intervention Group
- Control Group (Sham Comparator): This group will receive an educational brochure about physical activity during pregnancy.
  Interventions: Behavioral: Educational Brochure

INTERVENTIONS:
Behavioral: mHealth Intervention Group — Access to the mobile health application with exercise plans and education
  Arms: mHealth Intervention Group
Behavioral: Educational Brochure — An evidence-based educational brochure with general information about the benefits of physical activity during pregnancy
  Arms: Control Group

SUMMARY:
The goal of this pilot project is to test the feasibility and potential efficacy of the evidence-based mHealth app (BumptUp) for improving physical activity and subsequent health outcomes (i.e. obesity, hypertension, insulin resistance) among pregnant and postpartum women in a rural community.

In order to accomplish this goal, feasibility of the intervention protocol will be tested by the assessment of recruitment (how many participants eligible per month), retention (% of women who complete the study protocol), adherence to intervention (% of women who utilize the app), and acceptability (survey and one-on-one exit interviews) during pregnancy and postpartum.

Potential efficacy will be determined by examining trends in data on physical activity levels (achieving the goal of 150 minutes per week of physical activity (surveys and accelerometry)) between groups. Other secondary outcomes will also be assessed: weight status, body composition, blood pressure, insulin resistance, fitness levels, mental health, and infant anthropometrics.

Clinical hypotheses:

1. The mHealth program will be feasible as evidenced by high rates of enrollment, retention, and adherence, moderate-to-high levels of satisfaction, and low participant burden.
2. The mHealth intervention will show promise towards improving physical activity levels and other secondary outcomes in pregnant and postpartum women in a rural community.

DETAILED DESCRIPTION:
After contact is established and eligibility confirmed, Participants (N=40) will be enrolled and baseline surveys will be conducted to collect information about lifestyle, mental health, and anxiety levels. Patient data for those participants who have agreed to be in the study and have specifically agreed on the consent form to allow the study team to pull data from their prenatal charts. The data being pulled from charts will include patient weights, vital signs, blood pressures, current complications, blood analytes, and glucose tolerance test results from each prenatal visit. After the baby is born, delivery reports will also be obtained in order to collect information on the delivery outcomes (gender, mode of delivery, complications, time in labor) and baby's anthropometric data (birthweight, birth length, head circumference).

Compensation will be in the form of Amazon gift cards (delivered electronically). There will be 4 time points where they take the online assessments. At each time point, they will also be mailed an Actigraph accelerometer to wear for one week. These will be sanitized and mailed or dropped off to avoid any contamination from the study team to participants. When the week is over, the study team will check in with participants and discuss a plan for pick up. They can leave outside for a study team member to pick up (contactless ) or they can mail it back (with provided return envelope).

Each participant will still receive a total of $160. They be recruited and consented online around 18-20 weeks. Assessments will occur at 4 timepoints: baseline assessments at 23-25 weeks gestation ($40), phone check at 30 weeks, second assessment/set of surveys at 35-37 weeks ($40), delivery outcomes obtained, 6 week postpartum surveys ($40), and 12 week postpartum surveys ($40).

Statistical Analyses:

Sample Size Determination: Sample size for this pilot study was determined based on previously performed physical activity interventions among pregnant women. The effect size (0.91) for the main outcome of physical activity was determined from looking at post-intervention physical activity data from Asci et al.83. With this effect size, it was determined using SAS software with a type I error rate of 0.05 that a sample size of 20 per group could detect this difference with 80% power, thus our sample size of 15 per group is justified for a pilot project.

Data Analyses:

Aim 1: To estimate the success and feasibility of recruitment methods, the number of people who will hear about the study via various methods (e.g. health care providers, health fairs, word-of-mouth) will be estimated. Then, the number of women who completed initial screening, the number of women who meet the eligibility criteria, the number of women who complete each of the assessments, the number of women randomized, and the number of women who adhere to the intervention will be determined. The exit interview data will be analyzed via standard content analyses for qualitative studies as previously described84 (and recently performed by our group). Aim 2: Although the investigators may not detect all between group differences because the investigators are proposing a pilot project, appropriate statistical tests will be performed in order to examine trends, and thus, promise for effect in the larger future trial. Normality of the distribution for each variable will be tested using Kolmogorov-Smirnov tests, and non-normally distributed data will be transformed as needed. The baseline characteristics of the two groups will be compared using t-tests or Chi square tests. The potential effect of the intervention on study outcomes will be explored using repeated measures ANOVAs (group x time). Specifically, physical activity data between groups will be compared from pre-post intervention. All data will be entered in Redcap data management system. Analyses will be conducted using SAS or other statistical software.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 18-44
* 2) Confirmed singleton viable pregnancy
* 3) English-Speaking (the app is currently only available in English)
* 4) Physician release to participate in exercise
* 5) Ownership of a smart phone
* 6) Plans to deliver at The Medical Center in Bowling Green, KY.

Exclusion Criteria:

* 1) Multiple gestation pregnancy
* 2) Inability to provide voluntary informed consent
* 3) Any medical condition (pregnancy-related or not) that would preclude exercise.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2020-11-28 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility during pregnancy | Pregnancy (23-25 weeks gestation)
  how many participants eligible and successfully recruited per month
Protocol retention | 12 weeks postpartum
  % of women who complete the study protocol
Adherence to intervention | Pregnancy (35-37 weeks pregnant)
  % of women who use the app daily
Adherence to intervention | Postpartum (12 weeks after delivery)
  % of women who use the app daily
Acceptability of Intervention | Postpartum (12 weeks after delivery)
  measured via exit interviews
Physical activity levels | Pregnancy (23-25 weeks gestation)
  Assess the potential efficacy of the intervention by examining physical activity levels through objective actigraph data
Physical activity levels | Pregnancy (35-37 weeks gestation)
  Assess the potential efficacy of the intervention by examining physical activity levels through objective actigraph data
Physical activity levels | Postpartum (12 weeks)
  Assess the potential efficacy of the intervention by examining physical activity levels through objective actigraph data
Physical activity levels | Postpartum (6 weeks)
  Assess the potential efficacy of the intervention by examining physical activity levels through Exercise Vital Sign Survey

SECONDARY OUTCOMES:
Maternal weight status | Pregnancy (23-25 weeks gestation)
  Body weight (lbs)
Maternal weight status | Pregnancy (35-37 weeks gestation)
  Body weight (lbs)
Maternal weight status | Postpartum (12 weeks post-delivery)
  Body weight (lbs)
Maternal blood pressure | Pregnancy (23-25 weeks gestation)
  Assessed by nurse at clinical visit using standardized clinical equipment
Maternal blood pressure | Pregnancy (35-37 weeks gestation)
  Assessed by nurse at clinical visit using standardized clinical equipment
Maternal blood pressure | Postpartum (6 weeks post-delivery)
  Assessed by nurse at clinical using standardized clinical equipment
Maternal insulin resistance | Pregnancy (24-29 weeks gestation)
  Oral Glucose Tolerance Test Results
Maternal endothelial dysfunction | Pregnancy (35-37 weeks gestation)
  Assessed with a rapid, non-invasive technique that records endothelium-mediated changes in the peripheral arterial tone signal via a pair of finger probes
Maternal postpartum depression | Postpartum (12 weeks post-delivery)
  Edinburgh postpartum depression survey
Maternal mood | Pregnancy (23-25 weeks gestation)
  Profile of Mood Survey
Maternal mood | Pregnancy (35-37 weeks gestation)
  Profile of Mood Survey
Maternal mood | Postpartum (6 weeks post-delivery)
  Profile of Mood Survey
Maternal mood | Postpartum (12 weeks post-delivery)
  Profile of Mood Survey
Mental Health | Pregnancy (23-25 weeks gestation)
  Center for Epidemiological Studies Depression Survey
Mental Health | Pregnancy (35-37 weeks gestation)
  Center for Epidemiological Studies Depression Survey
Mental Health | Postpartum (6 weeks post-delivery)
  Center for Epidemiological Studies Depression Survey
Mental Health | Postpartum (12 weeks post-delivery)
  Center for Epidemiological Studies Depression Survey
Infant birthweight | At time of delivery
  Collected at delivery by trained nursing staff

CONTACTS AND LOCATIONS:
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No